CLINICAL TRIAL: NCT04021277
Title: Phase I Trial of the Combination of PS101-Mediated Acoustic Cluster Therapy (ACT) With Chemotherapy for Treatment of Liver Metastasis In Patients With Solid Tumours With an Expansion Cohort in Metastatic Colorectal And Pancreatic Cancer
Brief Title: PS101-mediated ACT With Chemotherapy in Liver Metastases From Cancer of Gastrointestinal Origin
Acronym: ACT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reason
Sponsor: EXACT Therapeutics AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PS101-01-2018; 2018-004609-16 (EudraCT Number)
Record Dates: First submitted 2019-07-03; First posted 2019-07-16 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor; Colorectal Cancer
Keywords: PS101-mediated ACT: the combination of PS101 with ultrasound; PS101-mediated ACT procedure: PS101 and ultrasound; ACT treatment: 3 × PS101-mediated ACT procedures
MeSH Terms: conditions — Colorectal Neoplasms | interventions — PS-101; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Part 1 is divided into two stages:
  Part 1a: 3+3 open label non-randomized design to evaluate two doses
  Part 1b: Single blind, randomized design to evaluate two doses
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and radiologist are blinded to treatment dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1a: ACT with chemotherapy in metastatic solid tumours (Experimental): 20 uL/kg or 40 uL/kg PS101 administered together with standard of care chemotherapy (FOLFOX or FOLFIRI) and ultrasound insonation over the targeted liver metastasis in patients with solid tumours
  Interventions: Drug: 20 uL/kg PS101; Drug: 40 uL/kg PS101; Device: Ultrasound
- Part 1b ACT with chemotherapy in metastatic CRC (Experimental): 20 uL/kg or 40 uL/kg PS101 administered together with standard of care chemotherapy (FOLFIRI) and ultrasound insonation over the targeted liver metastasis in patients with metastatic colorectal cancer
  Interventions: Drug: 20 uL/kg PS101; Drug: 40 uL/kg PS101; Device: Ultrasound

INTERVENTIONS:
Drug: 20 uL/kg PS101 — 20 uL/kg PS101 and chemotherapy given for 4 cycles over 6 weeks
Drug: 40 uL/kg PS101 — 40 uL/kg PS101 and chemotherapy given for 4 cycles over 6 weeks
Device: Ultrasound — Ultrasound activation and enhancement

SUMMARY:
Part 1: This clinical study will first test the safety and initial effect on the tumour of PS101-mediated ACT when given in combination with standard of care chemotherapy in patients with liver metastases (initially those with any solid tumors and then further in patients just with colorectal cancer [CRC]) in order to identify the recommended dose and schedule of PS101-mediated ACT that can be taken forward for further testing.

Part 2: Based on the Part 1 results, another part in patients with liver metastases from CRC and pancreatic cancer (if indicated) may take place following a substantial protocol amendment.

This record will focus on Part 1 of the study only and will be updated if Part 2 occurs.

DETAILED DESCRIPTION:
The suboptimal delivery of an anticancer agent to the target cancer cells represent a significant problem in many solid tumours, as it compromises the effectiveness of established therapeutics. If the amount of drug that reached any tumour could be increased without changing the amount administered systemically, it should be possible to increase the effectiveness of the treatment without adding to systemic toxicity.

PS101-mediated ACT involves the use of an experimental drug and an experimental device in patients with colon/rectal cancer that has spread to the liver and is given in combination with standard of care chemotherapy. The experimental drug, called PS101, is a liquid containing a mixture of positively and negatively charged microbubbles and microdroplets. It is injected into a vein (blood vessel) and from there follows the blood flow around the body to where the cancerous tumours are found. PS101 is given at the same time as a special type of ultrasound (performed using an ultrasound device) at the place in the liver where the cancerous tumour is found. The combination of PS101 and ultrasound is called Acoustic Cluster Therapy (ACT).

PS101-mediated ACT can potentially increase the uptake of an anticancer agent over the ultrasound targeted area. The preclinical development of PS101-mediated ACT suggests that this therapy may be of meaningful benefit while significant additional toxicity is not anticipated.

ELIGIBILITY:
MAIN INCLUSION CRITERIA

Providing informed consent and able to co-operate with the study requirements.

Diagnosis of any advanced solid tumour with liver metastases suitable for FOLFOX or FOLFIRI chemotherapy (Part 1a) / Diagnosis of any metastatic CRC with liver metastases suitable for FOLFIRI chemotherapy (Part 1b) .

At least two distinct target liver metastases (visible on computed tomography (CT)/magnetic resonance imaging (MRI) and of a suitable size), one being suitable for ultrasound and suitably spaced apart.

Eastern Co-operative Oncology performance status of 0 or 1 and with a predicted meaningful survival of at least 6 months.

. Suitable laboratory test results to receive chemotherapy.

Females who are not pregnant or lactating; males and females willing to follow contraceptive requirements.

Able to receive CT/MRI contrast agents.

MAIN EXCLUSION CRITERIA

Liver metastases suitable for immediate resection (and therefore neoadjuvant therapy unnecessary) or planned to be treated with radio-frequency ablation or other local therapies.

Liver radiotherapy in the last 2 months.

Use of tyrosine kinase inhibitors or monoclonal antibodies that are known to target angiogenesis receptors and/or their ligands.

Persistent, unresolved National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) Version 5.0 Grade 2 or higher drug-related toxicity (except alopecia, erectile dysfunction, hot flashes, decreased libido) following previous treatment.

Grade 2 or greater sensory/motor neuropathy.

Inadequate recovery from any prior surgical procedure or major surgical procedure in the last 4 weeks

Serious/symptomatic active infection, or infection requiring antibiotics in the last 7 days, active cholangitis, disease requiring metal biliary stent(s), HIV infection, bleeding diathesis or other medical or psychiatric condition that might interfere with the patient's participation in the trial or results.

Hypersensitivity to any of the components of PS101 (e.g. eggs or egg products).

Hypersensitivity to FOLFOX or FOLFIRI, or previously having to discontinue either due to adverse events.

Participation in any other clinical trials involving therapeutic agents in the last 4 weeks.

History of QT prolongation, clinically significant ventricular tachycardia, ventricular fibrillation, heart block, myocardial infarction within 6 months, congestive heart failure New York Heart Association Class III or IV, unstable angina or any relevant clinical history, signs or symptoms suggestive of clinically significant, uncontrolled cardiovascular or pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: DLTs (Part 1a only) | 4 weeks from the first ACT treatment in each patient
  Proportion of patients with DLTs related to administration of PS101 IV bolus injection alone (without chemotherapy) or due to the addition of PS101 to FOLFOX or FOLFIRI
Number of patients with adverse events | From informed consent to 12 weeks from study start
  Adverse events are summarised in the adverse event section. An overall summary will be presented here
Number of patients with adverse device effects | From the first PS101-mediated ACT procedure to 12 weeks from study start
  Number of patients with any AE related to the use of an Investigational Medical Device.

SECONDARY OUTCOMES:
Preliminary anti-tumor activity at Week 8 | Baseline to Week 8
  Change from baseline in maximum tumor diameter and volume in liver metastases
Best overall response (Part 1b only) | Baseline to 24 weeks
  Best overall response based on CR, PR, SD, PR according to RECIST Version 1.1

CONTACTS AND LOCATIONS:
Locations (4):
- Oslo University Hospital HF, Oslo, Norway
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan CH, Ho YJ, Lin CW, Wu N, Chiang PH, Yeh CK. State-of-the-art of ultrasound-triggered drug delivery from ultrasound-responsive drug carriers. Expert Opin Drug Deliv. 2022 Aug;19(8):997-1009. doi: 10.1080/17425247.2022.2110585. Epub 2022 Aug 10. PMID 35930441